CLINICAL TRIAL: NCT07227207
Title: A Phase 1/2, Open-Label, Multi-Center, Dose Escalation, Dose Expansion, and Single Repeat Dose Study of TSRA-196 in Adults With the PiZZ Genotype Who Have Lung and/or Liver Disease Associated With Severe Alpha-1 Antitrypsin Deficiency
Brief Title: A Study of TSRA-196 in Adults With PiZZ Alpha-1 Antitrypsin Deficiency (AATD)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tessera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSRA196-AAT-201
Record Dates: First submitted 2025-11-03; First posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Alpha-1 Antitrypsin Deficiency (AATD)
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TSRA-196 Drug Product (Experimental)
  Interventions: Drug: TSRA-196

INTERVENTIONS:
Drug: TSRA-196 — TSRA-196 is an in-vivo genome editing product formulated in lipid nanoparticles (LNPs) for the treatment of patients with alpha-1 antitrypsin deficiency (AATD), via intravenous (IV) infusion

SUMMARY:
This is a Phase 1/2, open-label, multi-center, dose escalation (Part 1), dose expansion (Part 2), and single repeat dose (Part 3) study to evaluate the safety, tolerability, efficacy, and PK/PD parameters of TSRA-196 in adults with the PiZZ genotype who have lung and/or liver disease associated with severe alpha-1 antitrypsin deficiency (AATD)

ELIGIBILITY:
Inclusion Criteria:

* Males or females who are 18 to 70 years of age, inclusive, at the time of signing the informed consent
* Body mass index of 18 to 37 kg/m2, inclusive
* Confirmed diagnosis of AATD and PiZZ genotype
* At least one previous measure of blood total AAT level <11 µmol/L
* Nonsmoker for at least 6 months before screening and must remain nonsmoking for the entire study duration
* Either AAT treatment-naïve or washed out of all investigational or approved treatments that modify AAT levels for 5 half-lives or at least 4 weeks, whichever is longer, before TSRA-196 administration

Parts 1A and 2A (AATD lung disease with no or minimal liver fibrosis)

* Clinically significant lung disease, defined as 1) evidence of emphysema or bronchiectasis by computed tomography or 2) DLCO <70% of the predicted value or 3) ppFEV1 <80%
* ppFEV1 ≥35%
* METAVIR fibrosis score F0 or F1 confirmed by liver biopsy at screening, or a liver stiffness measure by FibroScan ≤7 kPa at screening
* FIB-4 index score ≤3.25 at screening
* ALT and/or AST <ULN at screening

Parts 1B and 2B (AATD liver disease with significant or severe liver fibrosis, with or without AATD lung disease)

* METAVIR fibrosis score F2 or F3 confirmed by liver biopsy at screening. A liver biopsy conducted within 12 months before screening is acceptable as a substitute.
* Liver stiffness measure by FibroScan >7 and ≤15 kPa at screening
* ALT and/or AST <2 x ULN at screening

Exclusion Criteria:

* Presence of genetic variation in SERPINA1 gene that may disrupt the function of TSRA-196, determined by screening genotyping
* History of liver disease unrelated to AATD, or history of or clinical signs of cirrhosis
* Significant lung disease not attributable to manifestations of AATD, as determined by the investigator
* History of one or more hospitalizations due to severe exacerbation of underlying lung disease during the year before screening or received IV antibiotics for treatment of a pulmonary infection within 6 months before screening
* Unstable AATD-related COPD, as determined by the investigator, or severe bronchiectasis
* Lung volume reduction surgery within 1 year before screening or plan to receive lung volume reduction surgery during the study period
* Documented chronic need for positive airway pressure therapy beyond nocturnal use
* Seropositive for human immunodeficiency virus (HIV) (HIV-1 or HIV-2)
* Seropositive for hepatitis B (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb] positive) with detectable HBV DNA
* Hepatitis C virus (HCV) RNA positive at screening (Parts 1A and 2A), or HCV RNA positive and/or HCV antibody positive at screening (Parts 1B and 2B)
* Has received an organ transplant or is on a waiting list for an organ transplant
* Prior treatment with gene therapy using viral vectors or intended to permanently change the patient's DNA
* Any investigational products within 30 days before dosing or plan to take an investigational product before the end of study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation): Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 1 Year
Part 2 (Dose Expansion): Proportion of participants who have serum levels of total alpha-1 antitrypsin (AAT) greater than or equal to Lower Limit of Normal (LLN) after TSRA-196 treatment | 1 Year
Part 3 (Single Repeated Dose): Proportion of participants who have serum levels of total alpha-1 antitrypsin (AAT) greater than or equal to Lower Limit of Normal (LLN) after a second dose of TSRA-196 | 1 Year

SECONDARY OUTCOMES:
Part 1 (Dose Escalation): Proportion of participants who have serum levels of total AAT greater than or equal to LLN after TSRA-196 treatment | 1 Year
Part 2 (Dose Expansion): Incidence of TEAEs and SAEs | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): Proportion of participants who have serum levels of total AAT greater than or equal to 11 μM after TSRA-196 treatment | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): Change in serum levels of total AAT from baseline over time | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): Incidence of Adverse Event of Special Interest (AESI) from day of dosing through end of study | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): Change over time in safety measures, including clinical laboratory parameters, vital signs, and ECG parameters | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): Pharmacokinetic (PK) parameter: Area under the blood concentration time curves (AUC) of TSRA-196 | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): PK parameter: Maximum observed blood concentration (Cmax) of TSRA-196 | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): PK parameter: Time to Cmax (tmax) of TSRA-196 | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): PK parameter: Half-life (t1/2) of TSRA-196 | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): PK parameter: Clearance (CL) of TSRA-196 | 1 Year
Part 1 (Dose Escalation) and Part 2 (Dose Expansion): PK parameter: The volume of distribution at terminal stage (Vz) of TSRA-196 | 1 Year